CLINICAL TRIAL: NCT04108351
Title: Development and Validation of a Driving Simulator for Evaluating the Residual Effects of Drugs on Driving Performance - Sensitivity Analysis Using Zopiclone As a Positive Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Collaborators: Nagoya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: DS-204-04
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2020-02

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zopiclone (Experimental)
  Interventions: Other: Road-tracking test; Other: Car-following test; Other: Harsh-braking test
- Placebo (Placebo Comparator)
  Interventions: Other: Road-tracking test; Other: Car-following test; Other: Harsh-braking test

INTERVENTIONS:
Other: Road-tracking test — Driving with simulator program for SDLP measurement
Other: Car-following test — Intervention Description: Driving with simulator program for DCV measurement
Other: Harsh-braking test — Driving with simulator program for BRT measurement

SUMMARY:
The purpose of this study is to confirm of assay sensitivity of Driving Simulator by positive control

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.5 and <25.0 kg/m^2 at screening inspection
* No visual impairment (enable to correct the vision with eyeglasses or contact lens)
* Receive a prior explanation on the study, able to accept its content, and capable to provide voluntary written consent for participation in this study
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History of drug and food allergy
* Hypersensitivity to zopiclone
* Inappropriate for enrollment in this study was judged by principal investigator or subinvestigator
* Other protocol defined inclusion criteria could apply

Ages: 21 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP) | 60 min

SECONDARY OUTCOMES:
Distance Coefficient of Variation (DCV) | 5 min
Brake Reaction Time (BRT) | 5 min

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (2):
- Japan (2):
  - Taisho Pharmaceutical Co., Ltd selected site, Fukuoka
  - The medical facility selected by Taisho Pharmaceutical Co., Ltd, Fukuoka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iwata M, Iwamoto K, Kambe D, Tachibana N, Ando M, Ozaki N. Development and validation of a driving simulator for evaluating the residual effects of drugs on driving performance - sensitivity analysis using zopiclone as a positive control: Study Protocol Clinical Trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Mar;99(12):e19395. doi: 10.1097/MD.0000000000019395. PMID 32195934